CLINICAL TRIAL: NCT01138033
Title: A Phase I Open-Label Dose Escalation Study of the Focal Adhesion Kinase Inhibitor, GSK2256098, in Subjects With Solid Tumors
Brief Title: Study of a Focal Adhesion Kinase Inhibitor in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113517
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: pharmacodynamics; cancer; focal adhesion kinase inhibitor; pharmacokinetics; solid tumors; Phase 1
MeSH Terms: conditions — Neoplasms | interventions — GSK2256098

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 (Experimental): Part 1 - dose escalation; starting dose 80 mg BID
  Interventions: Drug: GSK2256098
- Part 2 (Experimental): Part 2 - Dose expansion phase of the study at the maximum tolerated dose and schedule identified in Part 1 in patients with tumors known to over express FAK
  Interventions: Drug: GSK2256098
- Part 3 (Experimental): Part 3 - Characterize the biologically active dose range by analysis of PD markers in skin, hair and in tumor tissue in subjects with solid tumors amendable to biopsy and know to over express FAK
  Interventions: Drug: GSK2256098
- Part 4 (Experimental): Part 4 - Explore further the safety, PK, tolerability and anti-tumor activity of GSK2256098 in subjects with relapsed glioblastoma multiforme (GBM).
  Interventions: Drug: GSK2256098
- Part 5 (Experimental): Part 5 will investigate the time course, the extent of an apparent change in the PK of GSK2256098 following repeated dosing, and screen for potential CYP3A induction as a possible mechanism of reduced systemic exposure of GSK2256098 at Day 15 and later time points.
  Interventions: Drug: GSK2256098

INTERVENTIONS:
Drug: GSK2256098 — GSK2256098 is a potent focal adhesion kinase inhibitor that will be administered orally as 20, 100 or 250 mg capsules. The starting dose in Part 1 is 80 mg twice daily. The dose will continue to be increased until the maximum tolerated dose is identified.

SUMMARY:
This study is a Phase I dose escalation study in subjects with solid tumors. Part 1 will identify the maximum tolerated dose (MTD) using a dose-escalation procedure. Following identification of the MTD, enrollment into Parts 2, 3, 4 and 5 may be concurrent. Part 2 will explore further the safety, PK, tolerability, and anti-tumor activity of GSK2256098 in subjects with tumors known to overexpress focal adhesion kinase (FAK). Part 3 will characterize the range of biologically effective doses by assessing pharmacodynamic (PD) markers in hair, skin and tumor tissue at doses that will not go lower than 80 mg or above the MTD dose levels tested during the Phase 1 dose escalation. Part 4 will explore further the safety, PK, tolerability and anti-tumor activity of GSK2256098 in subjects with relapsed glioblastoma multiforme (GBM). The primary objective of this study is to determine the safety, tolerability, and MTD of GSK2256098. Secondary objectives are to characterize the pharmacokinetics (PK) of GSK2256098; to identify a range of biologically active doses; to explore the anti-tumor activity of GSK2256098, and to explore relationships between GSK2256098 PK, PD and clinical endpoints. Part 5 will investigate the time course, the extent of an apparent change in the PK of GSK2256098 following repeated dosing, and screen for potential CYP3A induction as a possible mechanism of reduced systemic exposure of GSK2256098 at Day 15 and later time points. The primary objective of this study is to determine the safety, tolerability, and MTD of GSK2256098.

DETAILED DESCRIPTION:
This study is a Phase I dose escalation study in subjects with solid tumors. Part 1 will identify the maximum tolerated dose (MTD) using a dose-escalation procedure. Following identification of the MTD, enrollment into Parts 2, 3, 4, and 5 may be concurrent. Part 2 will explore further the safety, PK, tolerability, and anti-tumor activity of GSK2256098 in subjects with tumors known to overexpress focal adhesion kinase (FAK). Part 3 will characterize the range of biologically effective doses by assessing pharmacodynamic (PD) markers in hair, skin and tumor tissue at doses that will not go lower than 80 mg or above the MTD dose levels tested during the Phase 1 dose escalation. Part 4 will explore further the safety, PK, tolerability and anti-tumor activity of GSK2256098 in subjects with relapsed glioblastoma multiforme (GBM). The primary objective of this study is to determine the safety, tolerability, and MTD of GSK2256098. Secondary objectives are to characterize the pharmacokinetics (PK) of GSK2256098; to identify a range of biologically active doses; to explore the anti-tumor activity of GSK2256098, and to explore relationships between GSK2256098 PK, PD and clinical endpoints.

Subjects with solid tumors will receive GSK2256098 orally without interruption on consecutive days. The planned starting dose in Part 1 will be a total daily dose of 160 mg administered as 80 mg twice daily (BID) during the repeat dose phase of the study. In the first cohort, administration of study drug will be initiated as a single dose (80 mg) on Day 1 that will be followed by collection of PK samples. Subjects may then begin repeat dosing (80 mg BID) on Day 2 following the collection of the 24-h PK sample. In subsequent cohorts, administration of study drug will be given as a single dose (half the total daily dose) on Day 1 followed by collection of PK samples. Subjects may begin repeat dosing on Day 2 following collection of the 24-h PK sample.

During dose escalation (Part 1), a modified accelerated dose titration design will be followed by a standard 3+3 dose escalation design until the MTD is established. After the MTD is established approximately 30 additional subjects with tumors reported to have FAK over-expression will be enrolled to further explore the safety, tolerability and clinical activity of GSK2256098 (Part 2). Additional cohorts below the MTD may be expanded to further explore and characterize the range of biologically effective doses (Part 3). Part 4 will further explore the safety, PK, tolerability and anti-tumor activity of GSK2256098 in subjects with relapsed glioblastoma multiforme (GBM). Part 5 will investigate the time course, the extent of an apparent change in the PK of GSK2256098 following repeated dosing, and screen for potential CYP3A induction as a possible mechanism of reduced systemic exposure of GSK2256098 at Day 15 and later time points. The primary objective of this study is to determine the safety, tolerability, and MTD of GSK2256098.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* 18 years old or older.
* Confirmed diagnosis of a solid tumor malignancy that is not responsive to accepted standard therapies or for which there is no standard or curative therapy. Subjects with malignancies related to HIV infection or organ transplantation are excluded.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group scale
* Able to swallow and retain oral medication
* A male is eligible to enter and participate in the study if he either:
* agrees to abstain from sexual intercourse from the first dose of study drug and until 21 days after last dose of study medication, or
* agrees to use a condom and occlusive cap (diaphragm or cervical/vault cap) with spermicidal foam/gel/film/cream/suppository from the first dose of study drug and until 21 days after last dose of study medication,
* or is surgically sterile. NOTE: Male subjects must use contraception to prevent pregnancy in a female partner and prevent exposure of any partner to semen by any means (refer to Section 8.1).
* A female is eligible to enroll in the study if she is of:
* Non-child bearing potential (i.e., physiologically incapable of becoming pregnant) including any woman who is characterized by at least one of the following:

oHas had a hysterectomy oHas had a bilateral oophorectomy (ovariectomy) oHas had a bilateral tubal ligation oIs post-menopausal (total cessation of menses for ≥ 1 year)

* Childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following from at least 2 weeks prior to the first dose of study drug and until 21 days after last dose of study medication:
* Use an intrauterine device (IUD) with a documented failure rate of less than 1% per year.
* Have intercourse only with a vasectomized partner who is sterile and is the sole sexual partner for that woman.
* Complete abstinence from sexual intercourse.
* Use double barrier contraception defined as condom with occlusive cap (diaphragm or cervical/vault cap) with spermicidal foam/gel/film/cream/suppository from the first dose of study drug and until 21 days after last dose of study medication.

NOTE: Oral contraceptives are not reliable due to potential for drug-drug interaction.

* Adequate organ system function
* Paraffin-embedded, archival tumor tissue available for testing. If archival tissue is available but it is not feasible to obtain within the screening period, subjects may enroll and enter the study prior to these specimens being received for analyses. In situations that archival tumor specimens are not available, (i.e. insufficient archival tumor specimens or a local hospital refuses to release a tissue block or specimen for the purposes of the study), only subjects for Part 1 would be eligible under such circumstances if there is documentation to explain why this tissue is not available

Inclusion Criteria Part 2 and Part 3

* Confirmed cancers of the breast, esophagus, ovary, head and neck, colon, rectum, stomach, liver, endometrium, cervix, oral epithelium, thyroid, lung, prostate, sarcoma and other tumors reported in medical literature to overexpress FAK that are not responsive to accepted standard therapies or for which there is no standard or curative therapy.
* Subjects enrolled in Part 3 must have solid tumors that are amenable to biopsy.

Inclusion Criteria Part 4

* Subjects with glioblastoma multiforme at first or second recurrence defined as one or two progressions as Grade 4 astrocytic tumor since original diagnosis of any grade glioma.
* Subjects with prior treatment with bevacizumab (approximately 10 evaluable subjects) and subjects without prior treatment with anti-angiogenic therapy (includes bevacizumab and VEGFR inhibitors) will be allowed to enroll (approximately 10 evaluable subjects). For subjects with prior bevacizumab treatment, they should have progressed while receiving bevacizumab as defined by the RANO criteria. [WEN PY, 2010]
* Recurrent or refractory disease must meet all of the following criteria:
* Received prior chemoradiotherapy that incorporated temozolomide
* Confirmed true progressive disease (rather than pseudoprogression) according to the proposed RANO criteria [Wen PY, 2010]
* Progressive disease occurring within the first 12 weeks after completion of chemoradiotherapy must be radiographically documented (i.e., new area of enhancement) as being clearly outside the radiation field or must be pathologically confirmed
* Progressive disease occurring at ≥ 12 weeks after completion of chemoradiotherapy should include at least one of the following: -New contrast-enhancing lesion on decreasing, stable, or increasing doses of corticosteroids (new contrast- enhancing nonmeasurable disease is permitted) OR
* Increase of 25% in the sum of the products of perpendicular diameters of the contrast-enhancing lesions compared to baseline (e.g., 1st postradiotherapy scan) or best response after initiation of therapy while on stable or increasing doses of corticosteroids OR
* Significant increase in T2/FLAIR nonenhancing lesion (for subjects receiving antiangiogenic therapy) compared to baseline (e.g., 1st postradiotherapy scan) or best response after initiation of therapy on stable, or increasing doses of corticosteroids OR
* Clear radiographic progression of nonmeasurable lesions NOTE: An increase in corticosteroid dose or clinical deterioration not attributable to concurrent medication or comorbid conditions alone is not sufficient to indicate progressive disease for the purpose of entry onto the study.
* Documented radiographic presence of at least one measurable or non-measurable lesion as defined by the RANO criteria [Wen PY, 2010]
* If recent resection or biopsy of tumor has taken place, then all of the following must apply:
* Planned first dose of GSK2256098 must be > 28 days after surgery (or > 7 days after core needle biopsy)
* Subject has recovered from the effects of surgery
* Subject has at least one non-measurable residual lesion following surgery as defined by the RANO criteria [WEN PY, 2010]

Exclusion Criteria:

* Use of an investigational anti-cancer drug within 28 days or 5 half-lives with a minimum duration of 10 days from prior therapy preceding the first dose of GSK2256098 OR Chemotherapy within the last 3 weeks (6 weeks for prior nitrosourea or mitomycin C) OR any major surgery, radiotherapy, or immunotherapy within the last 4 weeks.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug. (To date there are no known approved drugs chemically related to GSK2256098.)
* Current use of a prohibited medication or requires any of these medications during treatment with GSK2256098 (Section 9.2).
* Current use of warfarin for therapeutic anticoagulation. NOTE: Low molecular weight heparin is permitted. PT/PTT must meet the inclusion criteria. .
* Presence of an active gastrointestinal disease or other condition known to interfere significantly with the absorption, distribution, metabolism, or excretion of drugs OR prior resection of small intestine.
* Unresolved toxicity greater than Grade 1 from previous anti-cancer therapy except alopecia.
* QTc interval > 450 msecs in males, 470 msec in women or congenital long QT syndrome. QTc calculation to be calculated by Fridericia formula. (Section 7.2.3)
* History of acute coronary syndromes (including unstable angina and myocardial infarction), atrial fibrillation, coronary angioplasty, or stenting within the past 24 weeks.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Symptomatic or untreated leptomeningeal or brain metastases. Subjects previously treated for these conditions who are asymptomatic and have not received corticosteroid and P450-inducing anti-epileptic medication for at least 2 months are permitted.
* Primary malignancy of the central nervous system.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Concurrent condition that in the Investigator's opinion would jeopardize compliance with the protocol.
* Nursing female.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice or kumquats, pummelos, exotic citrus fruit (i.e., star fruit, bitter melon), grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Any serious and/or unstable pre-existing medical, psychiatric or other condition (including lab abnormalities) that could interfere with subject safety or obtaining informed consent.

Additional Exclusion Criteria - Part 4 only:

- Subjects with >/=Grade 1 intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-07-27 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2015-12-21 (Actual)

PRIMARY OUTCOMES:
To evaluate the Maximum tolerated dose, identify the recommended Phase 2 dose(s), dose limiting toxicities, safety and tolerability of GSK2256098 given orally on consecutive days. | Until disease progression

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of GSK2256098 in blood after single- and repeat-dose administration | Until disease progression
To identify a range of biologically active doses | Until disease progression
To explore anti-tumor activity after treatment with GSK2256098 | Until disease progression
To explore relationships between GSK2256098 PK, PD and clinical endpoints | Until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Australia (2):
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- France (2):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Villejuif
- United Kingdom (4):
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Brown NF, Williams M, Arkenau HT, Fleming RA, Tolson J, Yan L, Zhang J, Singh R, Auger KR, Lenox L, Cox D, Lewis Y, Plisson C, Searle G, Saleem A, Blagden S, Mulholland P. A study of the focal adhesion kinase inhibitor GSK2256098 in patients with recurrent glioblastoma with evaluation of tumor penetration of [11C]GSK2256098. Neuro Oncol. 2018 Nov 12;20(12):1634-1642. doi: 10.1093/neuonc/noy078. PMID 29788497
- See also: Results for study 113517 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113517?search=study&search_terms=113517#rs